CLINICAL TRIAL: NCT06997068
Title: Decentralized Pilot Study of Triple Oral Metronomic Chemotherapy for Patients With Recurrent/Metastatic Oral Cavity Cancer in a Rural Midwest United States Population
Brief Title: Methotrexate, Erlotinib, and Celecoxib for the Treatment of Recurrent/Metastatic Oral Cavity Cancer in a Rural Midwest United States Population
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC240701; NCI-2025-03640 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-009083 (Other: Mayo Clinic Institutional Review Board); MC240701 (Other: Mayo Clinic)
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Oral Cavity Carcinoma; Recurrent Oral Cavity Carcinoma; Stage IVC Lip and Oral Cavity Cancer AJCC v8
MeSH Terms: conditions — Mouth Neoplasms | interventions — Celecoxib; Erlotinib Hydrochloride; X-Rays; Interviews as Topic; Methotrexate; merphos

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (methotrexate, erlotinib, celecoxib) (Experimental): Patients receive methotrexate PO on days 1, 8, 15, and 22 of each cycle, erlotinib PO QD on days 1-28 of each cycle, and celecoxib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo SOC imaging scans throughout the trial.
  Interventions: Drug: Celecoxib; Drug: Erlotinib Hydrochloride; Procedure: Imaging Procedure; Other: Interview; Drug: Methotrexate; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Celecoxib — Given PO
  Other Names: Benzenesulfonamide, 4-[5-(4-methylphenyl)-3-(trifluoromethyl)-1H-pyrazol-1-yl]-; Celebrex; Elyxyb; Onsenal; SC-58635; YM 177
Drug: Erlotinib Hydrochloride — Given PO
  Other Names: CP 358; CP-358; Cp-358,774; CP358; OSI 774; OSI-774; OSI774; Tarceva
Procedure: Imaging Procedure — Undergo SOC imaging scans
  Other Names: Diagnostic Imaging Technique; Image Type; Imaging; Imaging (procedure); Imaging Procedures; Imaging Technique; imaging type; IMAGING_METHOD; imaging_type; Medical Imaging; Type of imaging
Other: Interview — Ancillary studies
Drug: Methotrexate — Given PO
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial gathers information on the feasibility, safety, and effect of giving methotrexate, erlotinib, and celecoxib in treating oral cavity cancer that has come back after a period of improvement (recurrent) or that has spread from where it first started (primary site) to other places in the body (metastatic) among rural Midwest patients. Methotrexate is in a class of medications called antimetabolites. It is also a type of antifolate. Methotrexate stops cells from using folic acid to make deoxyribonucleic acid and may kill tumor cells. Erlotinib is in a class of medications called kinase inhibitors. It works by blocking the action of a protein called EGFR that signals tumor cells to multiply. This helps slow or stop the spread of tumor cells. Celecoxib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving the combination of methotrexate, erlotinib, and celecoxib may be feasible, safe, and effective in treating rural Midwest patients with recurrent/metastatic oral cavity cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically confirmed diagnosis of relapsed/metastatic oral cavity cancer
* Measurable or non-measurable disease is allowed

  * Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
  * Non-measurable disease

    * NOTE: Other nonmeasurable lesions include clinically evident lesions not well visualized on imaging [e.g., oral cavity mass readily seen on physical exam but obscured on computed tomography (CT)], dermal metastases, and bone metastases
* Prior treatment:

  * One of the following must be true:

    * Received standard 1st-line immunotherapy or chemo-immunotherapy OR
    * Unable to receive or refuse 1st-line therapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0, 1 or 2
* Hemoglobin ≥ 9.0 g/dL (obtained 15 days prior to registration)
* Absolute neutrophil count (ANC) ≥ 1500/mm^3 (obtained 15 days prior to registration)
* Platelet count ≥ 100,000/mm^3 (obtained 15 days prior to registration)
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (obtained 15 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤ 3 x ULN (≤ 5 x ULN for patients with liver involvement) (obtained 15 days prior to registration)
* Prothrombin time (PT)/international normalized ratio (INR)/activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN OR if patient is receiving anticoagulant therapy and INR or aPTT is within target range of therapy (obtained 15 days prior to registration)
* Calculated creatinine clearance ≥ 45 ml/min per Chronic-Kidney Disease-Epidemiology (CKD-EPI) Creatinine Equation (obtained 15 days prior to registration)
* Estimated creatinine clearance (Clcr) by the CKD-EPI Creatinine Equation (per National Kidney Foundation) (obtained 15 days prior to registration)
* Negative pregnancy test done ≤ 8 days prior to registration, for persons of childbearing potential only
* Provide written informed consent
* Ability to complete questionnaire(s) by themselves or with assistance
* Ability to swallow pills
* Willing and able to adhere with the protocol schedule for the duration of the study including undergoing treatment, attending scheduled visits, and examinations

Exclusion Criteria:

* Any of the following because this study involves an investigational agent, the genotoxic, mutagenic, and teratogenic effects of which on the developing fetus and newborn are unknown

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential and persons able to father a child who are unwilling to employ adequate contraception
* Uncontrolled intercurrent illness including, but not limited to:

  * Myocardial infarction ≤ 6 months prior to registration
  * New York Heart Association (NYHA) class III or IV heart failure
  * Corrected QT interval (QTc) prolongation more than 440 ms in males and 460 ms in females
  * Uncontrolled dysrhythmias or poorly controlled angina
  * History of serious ventricular arrhythmia [ventricular tachycardia (VT) or ventricular flutter (VF)] and/or factors that predispose to arrhythmia (e.g., heart failure, hypokalemia, family history of long QT syndrome)
  * Ongoing or active infection requiring systemic treatment
  * Active gastrointestinal bleeding
  * Psychiatric illness/social situations that would limit compliance with study requirements
* Immunocompromised patients and patients known to be HIV positive and currently receiving antiretroviral therapy

  * NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Known hepatitis

  * Exception: For patients with evidence of chronic hepatitis B virus infection the hepatitis B (HepB) viral load must be undetectable on suppressive therapy, if indicated, to be eligible
  * Exception: Patients with a history of hepatitis C virus infection must have been treated and cured. Patients with hepatitis C virus (HCV) infection who are currently on treatment are eligible if they have an undetectable HCV viral load
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy requiring therapy such as radiation, chemotherapy, or immunotherapy. Patients on hormonal therapy for treated breast or prostate cancer are permitted if they meet other eligibility criteria

  * NOTE: Patients with secondary malignancy with life expectancy ≥ 2 years are eligible
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Rates of provider referral and patient enrollment (Feasibility) | Up to 2 years
  Will capture the provider/patient reasons for declining trial participation. All information will be described descriptively. Categorical variables will be described with frequencies and percentages. Continuous variables will be described with means, medians, standard deviations, etc.
Rate of retention (Feasibility) | Up to 2 years
  Will capture the reasons for trial drop-out and assess adherence to treatment and reasons for deviation through qualitative and semiquantitative means. All information will be described descriptively. Categorical variables will be described with frequencies and percentages. Continuous variables will be described with means, medians, standard deviations, etc.
Rate of conversion from virtual to in-person visits (Feasibility) | Up to 2 years
  Will capture the provider/patient reasons for the switch and quantify the out-of-pocket costs of in-person and virtual visits. All the information will be described descriptively. Categorical variables will be described with frequencies and percentages. Continuous variables will be described with means, medians, standard deviations, etc.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 30 days after completion of study treatment
  The maximum grade for each type of adverse event will be recorded for each patient, assessed per Common Terminology Criteria in Adverse Events (CTCAE) version 5.0.
Objective response rate | Up to 3 years
  Defined as the proportion of participants who have a partial response or complete response, as assessed using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Progression-free survival | Up to 3 years
  Defined as the time from study entry until the first of either disease progression or death from any cause.
Overall survival | Up to 3 years
  Defined as the time from study entry until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Katharine A. Price, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials